CLINICAL TRIAL: NCT03189654
Title: Noninvasive Ventilation Therapy for the Treatment of Pleural Effusion in Patients With Heart Failure
Status: Completed | Type: Observational
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Collaborators: ResMed GmbH & Co KG (Unknown)
Responsible Party: Principal Investigator, Thomas Bitter, Senior physician, Heart and Diabetes Center North-Rhine Westfalia
Other Study IDs: HDZNRW-KA_010_TB
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Pleural Effusion; Heart Failure
MeSH Terms: conditions — Pleural Effusion; Heart Failure | interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment group: Non-invasive ventilation after pleurocentesis
  Interventions: Device: Non-invasive ventilation
- Control group: Oxygen Administration via nasal tube

INTERVENTIONS:
Device: Non-invasive ventilation — Non-invasive Ventilation for a Minimum of 8 h per day after pleurocentesis
  Groups: Treatment group

SUMMARY:
There are no investigations so far whether an application of positive pressure during non-invasive ventilation might be a therapeutic option for transudative pleural effusion in patients with heart failure. In view of the pathophysiological process with pleural effusion resulting from an increase in intravascular hydrostatic pressure, non-invasive ventilation might provide an improvement.

The aim of the present study is to investigate whether an additional non-invasive ventilation therapy leads to an improved suppression of pleural effusion in heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to our hospital on a routine or emergency basis
* Patients with heart failure according to the current ESC guidelines and chronic pleural effusion with clinical indication for pleurocentesis
* Non-invasively determined cardiac index of < 2.5 l/min/m²
* BNP > 300 pg/ml
* Transudative pleural effusion according to Light criteria
* Effective pleurocentesis with residual effusion on the side affected of < 500 ml
* Tolerance of non-invasive ventilation without subjective or objective hemodynamic impairment as verified during a test ventilation
* No change in drug or other therapy for the duration of the study (5 days)

Exclusion Criteria:

* Psychological or neurological concomitant disease making an informed consent impossible
* Pregnancy
* Pneumothorax or pneumomediastinum
* Pathologically low blood pressure, particularly associated with intravascular volume depletion
* Liquor discharge, recent head surgery or trauma
* Severe bullous lung disease
* Dehydration
* Current ventilation therapy
* Bilateral pleural effusion > 500 ml at the time of enrolment
* Exudative pleural effusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with decompensated heart failure and pleural effusion
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Amount of pleural effusion | 5 days

SECONDARY OUTCOMES:
nt-Pro-BNP | 5 days
Cardiac output | 5 days
NYHA class | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bitter, MD, Principal Investigator — Heart and Diabetes Center North Rhine-Westphalia
Locations (1):
- Clinic for Cardiology, Herz- und Diabeteszentrum NRW, Ruhr-Universität Bochum, Bad Oeynhausen, Germany

IPD SHARING:
Plan to Share IPD: No